CLINICAL TRIAL: NCT01290159
Title: Preliminary Study of Identifying the Tolerance to Heat by a Novel Biomarker of Oxidative Stress
Brief Title: The Development Of A Novel Biomarker For Early Identification Of The Individual's State Of Tolerance To Heat
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Yoram Epstein, Heller institue, Sheba Medical Center, Sheba Medical Center
Other Study IDs: SHEBA-10-8150-CM-CTIL
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Heat Stroke; Healthy
Keywords: tolerance to heat
MeSH Terms: conditions — Heat Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- post heat stroke heat tolerant
  Interventions: Other: heat tolerance test (HTT)
- post heat stroke heat intolerant
  Interventions: Other: heat tolerance test (HTT)
- healthy controls
  Interventions: Other: heat tolerance test (HTT)

INTERVENTIONS:
Other: heat tolerance test (HTT) — An exercise-heat test,which consists of 120 min exposure to walking on a treadmill (5km/h; 2% grade) under conditions of 40oC and 50% rh.
  Other Names: heat strain

SUMMARY:
Today, the level of tolerance to heat is based on physiological strain indices, with no correlates to any relevant biomarker. We hypothesize that oxidative stress (OS) and the formation of reactive oxygen and nitrogen species (ROS, RNS), which are part of the underling pathophysiology related to hyperthermia, can be used to identify tolerance/intolerance to heat. The aim of the present project is to develop a simple assay, based on specific designed sensitive biomarkers of OS that can be detected in a small blood sample, and to possibly correlate each individual's state of tolerance to heat to the level of OS. These biomarkers specially designed and synthesized to form a novel probe (not present as such in biological organs). The method will be based on the incubation of the suggested biomarkers with the patient's blood sample and the measurement of the level and type of oxidative alteration of the markers. For this goal, post heat stroke patients, with different levels of tolerance to heat and subjects during a process of acclimation to heat will be studied. Such a method will add to our ability to better determine the level of tolerance to heat and not rely only on the measurements of temperature and heart rate during an exercise-heat stress.

ELIGIBILITY:
Inclusion Criteria:

for study group: post heat stroke subjects. for control group: healthy subjects matched by age to study group

Exclusion Criteria:

for control group: any prior heat illness, Diabetes, heart failure, high blood pressure (SBP >140mmHg), any febrile illness within the last two weeks prior to testing.

for study group: Diabetes, heart failure, high blood pressure (SBP >140mmHg), any febrile illness within the last two weeks prior to testing

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young (18-28 years old) post heat stroke subjects, and matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Epstein, PhD, Study Director — Heller Institute of Medical Research, Sheba Medical Center, Tel Hashomer; Amit Druyan, MD, Principal Investigator — Heller Institute of Medical Research, Sheba Medical Center
Locations (1):
- Heller Institute of Medical Research, Sheba Medical Center, Tel Litwinsky, Israel